CLINICAL TRIAL: NCT04326621
Title: Effectiveness of Pressure Release Technique in Patients With Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Gema Serrano-Hernanz, PhD, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Geserraher
Record Dates: First submitted 2020-03-19; First posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRT group (Experimental): pressure Release Technique and exercises
  Interventions: Other: Pressure Release Technique (PRT); Other: Control
- Exercises group (Active Comparator): Only exercises
  Interventions: Other: Pressure Release Technique (PRT); Other: Control

INTERVENTIONS:
Other: Pressure Release Technique (PRT) — A pressure applied on muscles trigger points with the finger of a physiotherapist and exercises
Other: Control — exercises

SUMMARY:
A Pressure Release Technique will be test in patient with low back pain compared to a sham

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain at least 6 months

Exclusion Criteria:

* hernia, neurologic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
VAS | immediately after treatment
  self reported pain
VAS | at 6 months
  self reported pain

IPD SHARING:
Plan to Share IPD: No